CLINICAL TRIAL: NCT05921409
Title: Development of a New Tool for the Diagnosis and Monitoring of Fibromyalgia "FIBROKIT"
Brief Title: Tool for Fibromyalgia Diagnosis and Effect of Extra Virgin Olive Oil
Acronym: FIBROKIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pronacera Therapeutics SL (Industry)
Collaborators: Centre for the Development of Industrial Technology, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IDI20210749; IDI-20210749 (Other Grant/Funding Number: Centre for the Development of Industrial Technology, Ministry of Science and Innovation)
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Olive oil; Nutrition; Mediterranean diet; Proteomics; Metagenomics; Microbiome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blinded, placebo controlled intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment (extra virgin olive oil) and placebo (olive oil) were packed in 50 ml opaque envelopes for patients masking. Letters A and B were assigned randomly to each treatment by an external person not participating in the study design or analysis for investigator masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MED DIET + AOVE (Experimental): A six-months nutritional intervention with a Mediterranean diet, daily supplemented with 50 ml of extra virgin olive oil. The intake of the oil was divided in the main meals and needed to be consumed without cooking.
  Interventions: Dietary Supplement: Extra Virgin Olive oil-supplemented Mediterranean Diet Intervention
- MED DIET + AO (Placebo Comparator): A six-months nutritional intervention with a Mediterranean diet, daily supplemented with 50 ml of olive oil. The intake of the oil was divided in the main meals and needed to be consumed without cooking.
  Interventions: Dietary Supplement: Olive oil-supplemented Mediterranean Diet Intervention

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive oil-supplemented Mediterranean Diet Intervention — This intervention (treatment) consist of taking Extra Virgin Olive Oil ("treatment" group made up of 103 patients and 22 healthy people) for 6 months, accompanied by Mediterranean diet-based menus. During this time, blood and stool samples were taken at different points: before the start of the intervention (T0), 3 months after the start (T1), at the end of the intervention in the sixth month (T2) and 6 months after leaving the study (TF). Hence, a total of 4 time points were taken for analysis: T0, T1, T2, TF. Additionally, and following these same time points, the physical and psychological health status of the participants will be evaluated using the SF-36 health questionnaire. Similarly, the course of the pathology in terms of the Fibromyalgia Impact Questionnaire (FIQ) score were recorded.
  Arms: MED DIET + AOVE
Dietary Supplement: Olive oil-supplemented Mediterranean Diet Intervention — This intervention (treatment) consist of taking Olive Oil ("placebo" group made up of 103 patients and 22 healthy people) for 6 months, accompanied by Mediterranean diet-based menus. During this time, blood and stool samples were taken at different points: before the start of the intervention (T0), 3 months after the start (T1), at the end of the intervention in the sixth month (T2) and 6 months after leaving the study (TF). Hence, a total of 4 time points were taken for analysis: T0, T1, T2, TF. Additionally, and following these same time points, the physical and psychological health status of the participants will be evaluated using the SF-36 health questionnaire. Similarly, the course of the pathology in terms of the Fibromyalgia Impact Questionnaire (FIQ) score were recorded.
  Arms: MED DIET + AO

SUMMARY:
PRONACERA THERAPEUTICS S.L. is a young biotechnological company focused on the development of genetic diagnostic tools and treatments for pathologies in different medical areas such as reproduction, fibromyalgia and rare diseases or with deficiencies in diagnosis, with the aim of helping to optimize health systems through improvement in terms and forms of diagnosis. Among the multiple lines of R+D+i that are currently being developed, the reproductive genomic line and endometrial functional molecular biology stand out. Specifically, it develops the design of markers and performs the genetic analysis of infertility focused on female endometrial tissue.

Fibromyalgia is a complex and common chronic pain disorder that affects 12 million Europeans. Along with other symptoms, fibromyalgia causes pain and general tenderness to touch. Currently this disease is diagnosed following the criteria established by the American College of Rheumatology (ACR) of a combination of relevant symptoms and the description of how the person feels. In other words, in practice it is a diagnosis by elimination. A patient suffering from fibromyalgia usually takes between 2 to 3 years to obtain the correct diagnosis. Health experts consider that fibromyalgia is a disease that is difficult to diagnose and that is associated with an expensive use of health system services.

With FIBROKIT, Pronacera aims to design and develop a new diagnostic and monitoring tool for fibromyalgia by designing a panel of specific plasma proteome and intestinal microbiome biomarkers and reducing the number of biological samples used. During the execution of this project, the company will have three leading research and innovation organizations in the sector (Helix BioS, CINUSA and CICbioGUNE) that will support Pronacera. FIBROKIT will have a cohort of 250 participants (206 patients and 44 healthy volunteers) to validate the diagnostic capacity of the tool and perform a robust biostatistical study.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic syndrome characterized mainly by the presence of widespread pain. This pain is usually accompanied by other alterations, both physically and psychologically, which, ultimately, seriously compromise people's quality of life, affecting their family, social and work environment and causing high social-sanitary costs. Although different factors such as an imbalance at the oxidative level or control of the inflammatory response have been studied, to date it is not known exactly what molecular alteration is responsible for the appearance and development of FM. This situation makes extremely difficult the search for a curative treatment and a specific and accurate laboratory diagnosis. The concept of FIBROKIT was born with the intention of solving both shortcomings. Thus, the main objective of this project is to fully design the panel of specific biomarkers to use in FIBROKIT. To achieve this great objective, three specific objectives have been set:

1. Design, based on new scientific evidence, the components of the molecular diagnostic panel focused on Peripheral Blood Mononuclear Cell-specific proteins, plasma proteome and intestinal microbiome biomarkers.
2. Increase the number of patients participating in the study to validate the diagnostic capacity of the kit with robust statistics.
3. Analytically validate the response of the new panel of molecular markers to the course of the pathology and its monitoring under a nutritional intervention with olive oil-supplemented mediterranean diet.

ELIGIBILITY:
Inclusion Criteria:

* Women between 40 and 59 years
* Do not carry out any type of guided and structured physical activity (detailed in the exclusion criteria)
* Follow a balanced diet in terms of the food source (fruits, vegetables, legumes, meat, fish, etc.).

Exclusion Criteria:

* Being outside the established age range (40-59) at the time of the start of the study
* Have practiced some type of structured or planned physical activity more than 2 times a week during the last month, such as:

  1. Go to collective classes of Yoga, Tai-Chi, Zumba, dance, gymnastics or similar
  2. Going for a walk, cycling, hiking or similar for 30 minutes or more than 10,000 steps per day
* Being underweight (BMI < 18.5) or type II or higher obesity (BMI > 34.9)
* Suffer and have been diagnosed with any of the following chronic pathologies:

any type of cancer

* Acquired Immunodeficiency Syndrome (AIDS)
* Inflammatory diseases (rheumatoid arthritis, osteoarthritis)
* Gastrointestinal diseases (Crohn's disease, ulcerative colitis)
* Cardiovascular diseases (atherosclerosis, cardiomyopathy, stroke)
* Autoimmune diseases (systemic lupus erythematosus, celiac disease, Hashimoto's thyroiditis, multiple sclerosis)
* Metabolic diseases (Type I and II Diabetes, Metabolic Syndrome)
* Having been under intensive pharmacological treatment (3 or more drugs daily) with non-steroidal anti-inflammatory drugs, corticosteroids, analgesics, or antidepressants during the month prior to the start of the study.
* Being under antioxidant supplementation (Glutathione, Coenzyme Q10, plant extracts, phenolic compounds)
* Consuming an amount greater than 12 g/day of alcohol, admitted in the context of the Mediterranean diet (Willett et al., 1995).

Smoking or consuming any type of narcotic substance (regardless of the amount and frequency)

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 250 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of Voltage dependent anion channel 1 protein (VDAC) | 0 weeks
  VDAC protein determination by western blot
Concentration of Voltage dependent anion channel 1 protein (VDAC) | 12 weeks
  VDAC protein determination by western blot
Concentration of Voltage dependent anion channel 1 protein (VDAC) | 24 weeks
  VDAC protein determination by western blot
Concentration of Voltage dependent anion channel 1 protein (VDAC) | 48 weeks
  VDAC protein determination by western blot
Concentration of Microtubule-associated proteins 1B light chain 3B (LC3B) | 0 weeks
  LC3B protein determination by western blot
Concentration of Microtubule-associated proteins 1B light chain 3B (LC3B) | 12 weeks
  LC3B protein determination by western blot
Microtubule-associated proteins 1B light chain 3B (LC3B) | 24 weeks
  LC3B protein determination by western blot
Concentration of Microtubule-associated proteins 1B light chain 3B (LC3B) | 48 weeks
  LC3B protein determination by western blot
Concentration of Plasma Proteins | 0 weeks
  Plasma proteome Analysis by label-free nano Liquid Chromatography coupled to tandem mass spectrometry after top-14 depletion
Concentration of Plasma Proteins | 12 weeks
  Plasma proteome Analysis by label-free nano Liquid Chromatography coupled to tandem mass spectrometry after top-14 depletion
Concentration of Plasma Proteins | 24 weeks
  Plasma proteome Analysis by label-free nano Liquid Chromatography coupled to tandem mass spectrometry after top-14 depletion
Concentration of Plasma Proteins | 48 weeks
  Plasma proteome Analysis by label-free nano Liquid Chromatography coupled to tandem mass spectrometry after top-14 depletion
Abundance of Bacteria from the Intestinal Microbiome | 0 weeks
  Fecal metagenomic analysis by amplicon sequencing of hypervariable region V3-V4 from RNA 16S bacterial gene
Abundance of Bacteria from the Intestinal Microbiome | 12 weeks
  Fecal metagenomic analysis by amplicon sequencing of hypervariable region V3-V4 from RNA 16S bacterial gene
Abundance of Bacteria from the Intestinal Microbiome | 24 weeks
  Fecal metagenomic analysis by amplicon sequencing of hypervariable region V3-V4 from RNA 16S bacterial gene
Abundance of Bacteria from the Intestinal Microbiome | 48 weeks
  Fecal metagenomic analysis by amplicon sequencing of hypervariable region V3-V4 from RNA 16S bacterial gene

SECONDARY OUTCOMES:
36-Item Short Form Health Survey (SF-36) Score | 0 weeks
  36-Item Short Form Health Survey score
36-Item Short Form Health Survey (SF-36) Score | 12 weeks
  36-Item Short Form Health Survey score
36-Item Short Form Health Survey (SF-36) Score | 24 weeks
  36-Item Short Form Health Survey score
36-Item Short Form Health Survey (SF-36) Score | 48 weeks
  36-Item Short Form Health Survey score
Fibromyalgia Impact Questionnaire (FIQ) Score | 0 weeks
  Fibromyalgia Impact Questionnaire (FIQ) score
Fibromyalgia Impact Questionnaire (FIQ) Score | 12 weeks
  Fibromyalgia Impact Questionnaire (FIQ) score
Fibromyalgia Impact Questionnaire (FIQ) Score | 24 weeks
  Fibromyalgia Impact Questionnaire (FIQ) score
Fibromyalgia Impact Questionnaire (FIQ) Score | 48 weeks
  Fibromyalgia Impact Questionnaire (FIQ) score

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Sánchez Alcázar, MD, Study Chair — Pablo de Olavide University, Seville (Spain)
Locations (1):
- Pronacera Therapeutics Laboratory, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Lara A, Moreno-Fernandez AM, Jimenez-Guerrero M, Diaz-Lopez C, De-Miguel M, Cotan D, Sanchez-Alcazar JA. Mitochondrial Imbalance as a New Approach to the Study of Fibromyalgia. Open Access Rheumatol. 2020 Aug 24;12:175-185. doi: 10.2147/OARRR.S257470. eCollection 2020. PMID 32922097
- [Background] Ramirez-Tejero JA, Martinez-Lara E, Rus A, Camacho MV, Del Moral ML, Siles E. Insight into the biological pathways underlying fibromyalgia by a proteomic approach. J Proteomics. 2018 Aug 30;186:47-55. doi: 10.1016/j.jprot.2018.07.009. Epub 2018 Jul 17. PMID 30030163
- [Background] Minerbi A, Fitzcharles MA. Gut microbiome: pertinence in fibromyalgia. Clin Exp Rheumatol. 2020 Jan-Feb;38 Suppl 123(1):99-104. Epub 2020 Feb 12. PMID 32116215
- [Background] Clos-Garcia M, Andres-Marin N, Fernandez-Eulate G, Abecia L, Lavin JL, van Liempd S, Cabrera D, Royo F, Valero A, Errazquin N, Vega MCG, Govillard L, Tackett MR, Tejada G, Gonzalez E, Anguita J, Bujanda L, Orcasitas AMC, Aransay AM, Maiz O, Lopez de Munain A, Falcon-Perez JM. Gut microbiome and serum metabolome analyses identify molecular biomarkers and altered glutamate metabolism in fibromyalgia. EBioMedicine. 2019 Aug;46:499-511. doi: 10.1016/j.ebiom.2019.07.031. Epub 2019 Jul 18. PMID 31327695
- [Derived] Duran-Gonzalez E, Ramirez-Tejero JA, Perez-Sanchez M, Morales-Torres C, Gomez-Morano R, Diaz-Lopez C, Martinez-Lara A, Cotan D. Fibromyalgia diagnosis from a multi-omics approach: a gut feeling. Front Microbiol. 2025 Oct 2;16:1641185. doi: 10.3389/fmicb.2025.1641185. eCollection 2025. PMID 41113645
- [Derived] Del Amo LL, Duran-Gonzalez E, Ramirez-Tejero JA, Martinez-Lara A, Cotan D. Study protocol for FIBROKIT: a new tool for fibromyalgia diagnosis and patient follow-up. Front Neurol. 2023 Nov 21;14:1286539. doi: 10.3389/fneur.2023.1286539. eCollection 2023. PMID 38073622